CLINICAL TRIAL: NCT01780506
Title: A Phase 3, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide Versus Elvitegravir/Cobicistat/Emtricitabine/ Tenofovir Disoproxil Fumarate in HIV-1 Positive, Antiretroviral Treatment-Naïve Adults
Brief Title: Study to Evaluate the Safety and Efficacy of E/C/F/TAF (Genvoya®) Versus E/C/F/TDF (Stribild®) in HIV-1 Positive, Antiretroviral Treatment-Naive Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-292-0104; 2012-004458-27 (EudraCT Number)
Record Dates: First submitted 2013-01-16; First posted 2013-01-31 (Estimated); Results first posted 2016-01-08 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-08

CONDITIONS: HIV; HIV Infections
Keywords: HIV; Treatment Naive; HIV 1 Infected; Female; Women
MeSH Terms: conditions — HIV Infections | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- E/C/F/TAF (Double-Blind Phase) (Experimental): E/C/F/TAF plus E/C/F/TDF placebo for 144 weeks
  Interventions: Drug: E/C/F/TAF; Drug: E/C/F/TDF Placebo
- E/C/F/TDF (Double-Blind Phase) (Active Comparator): E/C/F/TDF plus E/C/F/TAF placebo for 144 weeks
  Interventions: Drug: E/C/F/TDF; Drug: E/C/F/TAF Placebo
- Open-Label Extension Phase (Experimental): After study unblinding, participants who complete 144 weeks of the study had the option to receive open-label E/C/F/TAF until commercially available, or until Gilead Sciences terminated the study in that country.
  Interventions: Drug: E/C/F/TAF

INTERVENTIONS:
Drug: E/C/F/TAF — 150/150/200/10 mg FDC tablet administered orally once daily
  Other Names: Genvoya®
  Arms: E/C/F/TAF (Double-Blind Phase); Open-Label Extension Phase
Drug: E/C/F/TDF — 150/150/200/300 mg FDC tablet administered orally once daily
  Other Names: Stribild®
  Arms: E/C/F/TDF (Double-Blind Phase)
Drug: E/C/F/TDF Placebo — Tablet administered orally once daily
  Arms: E/C/F/TAF (Double-Blind Phase)
Drug: E/C/F/TAF Placebo — Tablet administered orally once daily
  Arms: E/C/F/TDF (Double-Blind Phase)

SUMMARY:
The primary objective of this study is to evaluate the efficacy of elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) fixed-dose combination (FDC) versus elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate (E/C/F/TDF) FDC in HIV-1 positive, antiretroviral treatment-naive adults.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* Plasma HIV-1 RNA levels ≥ 1,000 copies/mL at screening
* No prior use of any approved or investigational antiretroviral drug for any length of time, except the use for pre-exposure prophylaxis (PREP) or post-exposure prophylaxis (PEP), up to 6 months prior to screening
* Screening genotype report must show sensitivity to elvitegravir, emtricitabine, tenofovir disoproxil fumarate (tenofovir DF)
* Normal electrocardiogram (ECG)
* Estimated glomerular filtration rate (eGFR) ≥ 50 mL/min according to the Cockcroft-Gault formula for creatinine clearance
* Hepatic transaminases (AST and ALT) ≤ 5 × upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Adequate hematologic function
* Serum amylase ≤ 5 × ULN
* Males and females of childbearing potential must agree to utilize highly effective contraception methods or be non-heterosexually active or practice sexual abstinence from screening throughout the duration of study treatment and for 30 days following the last dose of study drug
* Females who utilize hormonal contraceptive as one of their birth control methods must have used the same method for at least three months prior to study dosing
* Females who have stopped menstruating for ≥ 12 months but do not have documentation of ovarian hormonal failure must have a serum follicle stimulating hormone (FSH) level at screening within the post-menopausal range based on the Central Laboratory reference range

Key Exclusion Criteria:

* A new acquired immunodeficiency syndrome (AIDS) defining condition diagnosed within the 30 days prior to screening
* Hepatitis B surface antigen (HBsAg) positive
* Hepatitis C antibody positive
* Individuals experiencing decompensated cirrhosis
* Females who are breastfeeding
* Positive serum pregnancy test
* Have an implanted defibrillator or pacemaker
* Current alcohol or substance use judged by the Investigator to potentially interfere with study compliance
* History of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, noninvasive cutaneous squamous carcinoma
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline
* Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the individual unsuitable for the study or unable to comply with dosing requirements
* Participation in any other clinical trial (including observational trials) without prior approval
* Individuals receiving ongoing therapy with drugs not to be used with elvitegravir, cobicistat, emtricitabine, tenofovir DF, and TAF or individuals with any known allergies to the excipients of E/C/F/TDF or E/C/F/TAF single-tablet regimen tablets

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 872 (Actual)
Dates: Start 2012-12-26 (Actual); Primary Completion 2014-08-26 (Actual); Study Completion 2017-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (117):
- United States (78):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Spectrum Medical Group, Phoenix, Arizona
  - Kaiser Permanente Los Angeles, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Peter J. Ruane, MD, Inc., Los Angeles, California
  - Anthony Mills MD Inc, Los Angeles, California
  - East Bay AIDS Center, Oakland, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - La Playa Medical Group and Clinical Research, San Diego, California
  - University of California, San Diego, San Diego, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Apex Research, LLC, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Dupont Circle Physicians Group, P.C., Washington D.C., District of Columbia
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - Capital Medical Associates, P.C., Washington D.C., District of Columbia
  - Gary Richmond, MD, PA, Inc., Fort Lauderdale, Florida
  - Midway Immunology & Research Center, LLC, Ft. Pierce, Florida
  - The Kinder Medical Group, Miami, Florida
  - AIDS Healthcare Foundation, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - IDOCF/ValuHealthMD, LLC, Orlando, Florida
  - Infectious Diseases Associates, Pensacola, Florida
  - The University of South Florida, Tampa, Florida
  - Infectious Disease Research Institute Inc., Tampa, Florida
  - St. Joseph's Comprenhensive Research Inisitute, Tampa, Florida
  - AIDS Research and Treatment Center of the Treasure Coast, Vero Beach, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Atlanta ID Group, PC, Atlanta, Georgia
  - Infectious Disease Specialist of Atlanta, Decatur, Georgia
  - Mercer University School of Medicine, Macon, Georgia
  - University of Hawaii - Hawaii Center for AIDS, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Ruth M. Rothstein CORE Center, Chicago, Illinois
  - Howard Brown Health Center, Chicago, Illinois
  - Institute of Human Virology, University of Maryland, Baltimore, Maryland
  - Community Research Initative, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Metrowest Medical Center, Framingham, Massachusetts
  - Baystate Infectious Diseases Clinical Research, Springfield, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Central West Clinical Research, Inc., St Louis, Missouri
  - Southampton Healthcare, Inc., St Louis, Missouri
  - ID Care, Hillsborough, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - Southwest C.A.R.E. Center, Santa Fe, New Mexico
  - Albany Medical College, Albany, New York
  - Upstate Infectious Diseases Associates, Albany, New York
  - New York Hospital Queens, Flushing, New York
  - North Shore University Hospital - Division of Infectious Diseases, Manhasset, New York
  - Mount Sinai School of Medicine, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Infectious Disease Consultants, PA, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - Summa Health Care Center, Akron, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of South Carolina School of Medicine, Columbia, South Carolina
  - Central Texas Clinical Research, Austin, Texas
  - St. Hope Foundation, Inc., Bellaire, Texas
  - Trinity Health and Wellness Center/AIDS Arms, Inc., Dallas, Texas
  - North Texas Infectious Diseases Consultants, Dallas, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Garcias' Family Health Group, Harlingen, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Gordon E. Crofoot, MD, PA, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Clinical Alliance for Research & Education - Infectious Diseases, LLC (CARE-ID), Annandale, Virginia
  - Peter Shalit, MD, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - Holdsworth House Medical Practice, Darlinghurst, New South Wales
  - Taylor Square Private Clinic, Darlington, New South Wales
  - East Sydney Doctors, Sydney, New South Wales
  - Albion Street Centre, Sydney, Southwest
  - Melbourne Sexual Health Clinic, Carlton, Victoria
- Austria (2):
  - DIAID, Department of Dermatology, Medical University Vienna, Vienna
  - Otto-Wagner-Spital, Sozialmedizinisches Zentrum Baumgartner Hoehe, Vienna
- Belgium (2):
  - Hôpital Erasme-ULB, Anderlecht, Brussels Capital
  - CHU Saint-Pierre University Hospital, Brussels
- Canada (8):
  - Spectrum Health, Vancouver, British Columbia
  - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - The Ottawa Hospital, Ottawa, Ontario
  - Maple Leaf Research, Toronto, Ontario
  - Clinique Medicale Du Quartier Latin, Montreal, Quebec
  - Clinique medicale l'Actuel, Montreal, Quebec
  - Clinique OPUS, Montreal, Quebec
  - Sunnybrook Health Science Center, Toronto
- Ospedale San Raffaele, Milan, Italy
- National Center for Global Health and Medicine AIDS Clinical Center, Shinjuku-ku, Tokyo, Japan
- HOPE Clinical Research, San Juan, Puerto Rico
- Spain (9):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - University Hospital Bellvitge, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela
- Switzerland (3):
  - Universitätsspital Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - University Hospital, Zurich, Zurich
- Thailand (6):
  - The HIV Netherland Australia Thailand, Thai Red Cross AIDS Research Center (The HIV-NAT), Bangkok
  - Ramathibodi Hospital, Mahidol University, Bangkok
  - Siriraj Hospital, Bangkok
  - Chiang Mai University, Chiang Mai
  - Khon Kaen University, Khon Kaen
  - Bamrasnaradura Infectious Diseases Institute, Nonthaburi
- Chelsea & Westminster Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Sax PE, Wohl D, Yin MT, Post F, DeJesus E, Saag M, Pozniak A, Thompson M, Podzamczer D, Molina JM, Oka S, Koenig E, Trottier B, Andrade-Villanueva J, Crofoot G, Custodio JM, Plummer A, Zhong L, Cao H, Martin H, Callebaut C, Cheng AK, Fordyce MW, McCallister S; GS-US-292-0104/0111 Study Team. Tenofovir alafenamide versus tenofovir disoproxil fumarate, coformulated with elvitegravir, cobicistat, and emtricitabine, for initial treatment of HIV-1 infection: two randomised, double-blind, phase 3, non-inferiority trials. Lancet. 2015 Jun 27;385(9987):2606-15. doi: 10.1016/S0140-6736(15)60616-X. Epub 2015 Apr 15. PMID 25890673
- [Result] Arribas JR, Thompson M, Sax PE, Haas B, McDonald C, Wohl DA, DeJesus E, Clarke AE, Guo S, Wang H, Callebaut C, Plummer A, Cheng A, Das M, McCallister S. Brief Report: Randomized, Double-Blind Comparison of Tenofovir Alafenamide (TAF) vs Tenofovir Disoproxil Fumarate (TDF), Each Coformulated With Elvitegravir, Cobicistat, and Emtricitabine (E/C/F) for Initial HIV-1 Treatment: Week 144 Results. J Acquir Immune Defic Syndr. 2017 Jun 1;75(2):211-218. doi: 10.1097/QAI.0000000000001350. PMID 28282300
- [Result] Margot N, Cox S, Das M, McCallister S, Miller MD, Callebaut C. Infrequent development of drug resistance in HIV-1-infected treatment-naive subjects after 96 weeks of treatment with elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide or elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate. Antivir Ther. 2017;22(5):443-446. doi: 10.3851/IMP3125. Epub 2017 Jan 11. PMID 28076335
- [Result] Margot NA, Kitrinos KM, Fordyce M, McCallister S, Miller MD, Callebaut C. Rare emergence of drug resistance in HIV-1 treatment-naive patients after 48 weeks of treatment with elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide. HIV Clin Trials. 2016 Mar;17(2):78-87. doi: 10.1080/15284336.2016.1142731. PMID 26892863
- [Result] Funderburg NT, McComsey GA, Kulkarni M, Bannerman T, Mantini J, Thornton B, Liu HC, Zhang Y, Song Q, Fang L, Dinoso J, Cheng A, McCallister S, Fordyce MW, Das M. Equivalent Decline in Inflammation Markers with Tenofovir Disoproxil Fumarate vs. Tenofovir Alafenamide. EBioMedicine. 2016 Nov;13:321-327. doi: 10.1016/j.ebiom.2016.10.009. Epub 2016 Oct 11. PMID 27742226
- [Result] Wohl D, Oka S, Clumeck N, Clarke A, Brinson C, Stephens J, Tashima K, Arribas JR, Rashbaum B, Cheret A, Brunetta J, Mussini C, Tebas P, Sax PE, Cheng A, Zhong L, Callebaut C, Das M, Fordyce M; GS-US-2,92-01040111 and Study Team. Brief Report: A Randomized, Double-Blind Comparison of Tenofovir Alafenamide Versus Tenofovir Disoproxil Fumarate, Each Coformulated With Elvitegravir, Cobicistat, and Emtricitabine for Initial HIV-1 Treatment: Week 96 Results. J Acquir Immune Defic Syndr. 2016 May 1;72(1):58-64. doi: 10.1097/QAI.0000000000000940. PMID 26829661
- [Result] Custodio JM, Garner W, Callebaut C, Fordyce M, Plummer A, Zhong L, et al. The Pharmacokinetics of Tenofovir and Tenofovir Diphosphate Following Administration of Tenofovir Alafenamide vs Tenofovir Disoproxil Fumarate [Oral Abstract #6]. The 16th International Workshop on Clinical Pharmacology of HIV & Hepatitis Therapy. Washington DC, USA, May 26-28, 2015.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, and Asia. The first participant was screened on 26 December 2012. The last study visit occurred on 06 September 2017.
Pre-assignment Details: 1105 participants were screened.
Groups:
- E/C/F/TAF: Double-Blind Phase: Elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) (150/150/200/10 mg) fixed-dose combination (FDC) tablet plus elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate (E/C/F/TDF) placebo tablet administered orally once daily for at least 144 weeks.
  Open-Label Extension Phase: After study unblinding, participants who completed 144 weeks of the study were given the option to receive open-label E/C/F/TAF (150/150/200/10 mg) FDC tablet until commercially available, or until Gilead Sciences terminated the study in that country.
- E/C/F/TDF: Double-Blind Phase: E/C/F/TDF (150/150/200/300 mg) FDC tablet plus E/C/F/TAF placebo tablet administered orally once daily for at least 144 weeks.
  Open-Label Extension Phase: After study unblinding, participants who completed 144 weeks of the study were given the option to receive open-label E/C/F/TAF (150/150/200/10 mg) FDC tablet until commercially available, or until Gilead Sciences terminated the study in that country.
Period: Double-Blind Phase
Arm/Group | E/C/F/TAF | E/C/F/TDF
Started | 438 | 434
Completed | 368 | 356
Not Completed | 70 | 78
Not completed — Randomized but not Treated | 3 | 2
Not completed — Adverse Event | 4 | 14
Not completed — Death | 1 | 2
Not completed — Pregnancy | 2 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Investigator's Discretion | 5 | 2
Not completed — Non-Compliance with Study Drug | 4 | 3
Not completed — Protocol Violation | 4 | 3
Not completed — Withdrew Consent | 23 | 24
Not completed — Lost to Follow-up | 23 | 26
Period: Open-Label Extension Phase
Arm/Group | E/C/F/TAF | E/C/F/TDF
Started | 90 (278 participants completed the Double-Blind Phase but did not enter the Open-Label Extension Phase) | 95 (261 participants completed the Double-Blind Phase but did not enter the Open-Label Extension Phase)
Completed | 90 | 94
Not Completed | 0 | 1
Not completed — Enrolled but not Treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug.
Groups:
- E/C/F/TAF: E/C/F/TAF (150/150/200/10 mg) FDC tablet plus E/C/F/TDF placebo tablet administered orally once daily for 144 weeks
- E/C/F/TDF: E/C/F/TDF (150/150/200/300 mg) FDC tablet plus E/C/F/TAF placebo tablet administered orally once daily for 144 weeks
- Total: Total of all reporting groups
Arm/Group | E/C/F/TAF | E/C/F/TDF | Total
Number analyzed (Participants) | 435 | 432 | 867
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (10.0) | 36 (10.5) | 35 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 56 | 127
  Male | 364 | 376 | 740
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60 | 70 | 130
  Not Hispanic or Latino | 375 | 362 | 737
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 5 | 9
  Asian | 76 | 77 | 153
  Black | 94 | 81 | 175
  Native Hawaiian or Pacific Islander | 1 | 3 | 4
  White | 250 | 255 | 505
  Other | 10 | 11 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 252 | 250 | 502
  Japan | 4 | 6 | 10
  United Kingdom | 1 | 5 | 6
  Thailand | 63 | 58 | 121
  Switzerland | 6 | 12 | 18
  Spain | 42 | 42 | 84
  Canada | 23 | 23 | 46
  Austria | 15 | 8 | 23
  Belgium | 7 | 7 | 14
  Italy | 3 | 6 | 9
  Australia | 19 | 15 | 34
HIV-1 RNA (log10 copies/mL) [Mean (Standard Deviation); unit: log10 copies/mL] | 4.55 (0.682) | 4.55 (0.674) | 4.55 (0.678)
HIV-1 RNA Category [Count of Participants; unit: Participants]
  ≤ 100,000 copies/mL | 331 | 336 | 667
  > 100,000 to ≤ 400,000 copies/mL | 79 | 72 | 151
  > 400,000 copies/mL | 25 | 24 | 49
CD4 Cell Count [Mean (Standard Deviation); unit: cells/µL] | 437 (223.7) | 426 (212.3) | 432 (218.0)
CD4 Cell Count Category [Count of Participants; unit: Participants]
  < 50 cells/µL | 10 | 12 | 22
  ≥ 50 to < 200 cells/µL | 48 | 41 | 89
  ≥ 200 to < 350 cells/µL | 103 | 111 | 214
  ≥ 350 to < 500 cells/µL | 122 | 135 | 257
  ≥ 500 cells/µL | 152 | 133 | 285
HIV Disease Status [Count of Participants; unit: Participants]
  Asymptomatic | 402 | 406 | 808
  Symptomatic HIV Infection | 23 | 15 | 38
  AIDS | 9 | 10 | 19
  Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Full Analysis Set: participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 435 | 432
percentage of participants | 93.1 | 92.8
Statistical Analysis 1: Comparison: E/C/F/TAF vs E/C/F/TDF; Test type: Non-Inferiority or Equivalence — Null hypothesis: the E/C/F/TAF group was ≥ 12% worse than the E/C/F/TDF group with respect to the percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48; alternative hypothesis: the E/C/F/TAF group was < 12% worse than the E/C/F/TDF group; p = 0.78, Cochran-Mantel-Haenszel — P-value was from the Cochran-Mantel-Haenszel (CMH) test stratified by baseline HIV-1 RNA (≤ 100,000 or > 100,000 copies/mL) and region (US vs ex-US); Difference in percentages = 0.5, 95.002% CI 2-sided [-3.0 to 4.0] — The difference in percentages and its 95.002% confidence interval (CI) were calculated based on the Mantel-Haenszel (MH) proportions adjusted by baseline HIV-1 RNA and region stratum

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Weeks 96 and 144
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Weeks 96 and 144 were analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Weeks 96 and 144
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 435 | 432
percentage of participants
  Week 96 | 89.2 | 88.2
  Week 144 | 86.9 | 83.1

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 20 Copies/mL at Weeks 48, 96, and 144
Description: The percentage of participants achieving HIV-1 RNA < 20 copies/mL at Weeks 48, 96, and 144 were analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Weeks 48, 96. and 144
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 435 | 432
percentage of participants
  Week 48 | 86.4 | 87.3
  Week 96 | 84.4 | 83.6
  Week 144 | 84.6 | 80.1

4. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with on-treatment data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 413 | 404
cells/µL | 235 (183.1) | 221 (178.9)

5. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 96
Time Frame: Baseline; Week 96
Population: Participants in the Full Analysis Set with on-treatment data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 395 | 384
cells/µL | 285 (203.0) | 271 (208.1)

6. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 144
Time Frame: Baseline; Week 144
Population: Participants in the Full Analysis Set with on-treatment data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 379 | 360
cells/µL | 323 (213.1) | 310 (207.2)

7. Secondary Outcome: Percent Change From Baseline in Hip Bone Mineral Density (BMD) at Week 48
Description: Hip BMD was assessed by dual energy x-ray absorptiometry (DXA) scan.
Time Frame: Baseline; Week 48
Population: Hip DXA Analysis Set: participants who were randomized and received at least 1 dose of study drugs and had nonmissing baseline hip BMD values. Participants were grouped according to the treatment they actually received. The missing-equals-excluded approach was used, where participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 404 | 394
percent change | -0.865 (3.2532) | -3.200 (3.1759)

8. Secondary Outcome: Percent Change From Baseline in Hip BMD at Week 96
Description: Hip BMD was assessed by DXA scan.
Time Frame: Baseline; Week 96
Population: Hip DXA Analysis Set. Participants were grouped according to the treatment they actually received. The missing-equals-excluded approach was used, where participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 375 | 365
percent change | -0.951 (3.8633) | -3.515 (3.9451)

9. Secondary Outcome: Percent Change From Baseline in Hip BMD at Week 144
Description: Hip BMD was assessed by DXA scan.
Time Frame: Baseline; Week 144
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 362 | 354
percent change | -0.826 (4.6786) | -3.475 (4.1551)

10. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 48
Description: Spine BMD was assessed by DXA scan.
Time Frame: Baseline; Week 48
Population: Spine DXA Analysis Set: participants who were randomized and received at least 1 dose of study drugs and had nonmissing baseline spine BMD values. Participants were grouped according to the treatment they actually received. The missing-equals-excluded approach was used, where participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 402 | 396
percent change | -1.337 (3.0715) | -2.956 (3.3524)

11. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 96
Description: Spine BMD was assessed by DXA scan.
Time Frame: Baseline; Week 96
Population: Spine DXA Analysis Set. Participants were grouped according to the treatment they actually received. The missing-equals-excluded approach was used, where participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 376 | 367
percent change | -0.907 (4.0039) | -3.053 (3.9539)

12. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 144
Description: Spine BMD was assessed by DXA scan.
Time Frame: Baseline; Week 144
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 369 | 352
percent change | -0.809 (4.5041) | -3.023 (4.3122)

13. Secondary Outcome: Change From Baseline in Serum Creatinine at Week 48
Time Frame: Baseline; Week 48
Population: Safety Analysis Set. The missing-equals-excluded approach was used, where participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 415 | 406
mg/dL | 0.08 (0.110) | 0.11 (0.116)

14. Secondary Outcome: Change From Baseline in Serum Creatinine at Week 96
Time Frame: Baseline; Week 96
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 398 | 386
mg/dL | 0.05 (0.109) | 0.07 (0.132)

15. Secondary Outcome: Change From Baseline in Serum Creatinine at Week 144
Time Frame: Baseline; Week 144
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 384 | 362
mg/dL | 0.04 (0.115) | 0.08 (0.133)

16. Secondary Outcome: Percentage of Participants Experiencing Treatment-emergent Proteinuria Through Week 48
Description: Grades 1 (mild), 2 (moderate), and 3 (severe) were the highest treatment-emergent postbaseline grades for urine protein using the dipstick method. The worst postbaseline value is presented for each participant.
Time Frame: Up to 48 weeks
Population: Participants in the Safety Analysis Set with at least 1 postbaseline urine protein value were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 434 | 431
percentage of participants
  Grade 1 | 25.8 | 32.3
  Grade 2 | 4.6 | 4.9
  Grade 3 | 0 | 0.2

17. Secondary Outcome: Percentage of Participants Experiencing Treatment-emergent Proteinuria Through Week 96
Description: as for outcome 16
Time Frame: Up to 96 weeks
Population: Participants in the Safety Analysis Set with at least 1 postbaseline urine protein value were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 434 | 431
percentage of participants
  Grade 1 | 28.8 | 33.9
  Grade 2 | 5.1 | 5.8
  Grade 3 | 0.2 | 0.2

18. Secondary Outcome: Percentage of Participants Experiencing Treatment-emergent Proteinuria Through Week 144
Description: as for outcome 16
Time Frame: Up to 144 weeks
Population: Participants in the Safety Analysis Set with at least 1 postbaseline urine protein value were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 434 | 431
percentage of participants
  Grade 1 | 31.3 | 37.1
  Grade 2 | 6.0 | 7.0
  Grade 3 | 0.2 | 0.2

19. Secondary Outcome: Percent Change From Baseline in Urine Retinol Binding Protein (RBP) to Creatinine Ratio at Week 48
Description: Urine RBP is a renal biomarker which is used to detect drug-induced kidney injury.
Time Frame: Baseline; Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 411 | 403
percent change | 6.9 [-23.3 to 42.1] | 51.2 [3.3 to 127.1]

20. Secondary Outcome: Percent Change From Baseline in Urine RBP to Creatinine Ratio at Week 96
Description: Urine RBP is a renal biomarker which is used to detect drug-induced kidney injury.
Time Frame: Baseline; Week 96
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 393 | 382
percent change | 11.3 [-20.3 to 61.5] | 75.0 [9.9 to 182.6]

21. Secondary Outcome: Percent Change From Baseline in Urine RBP to Creatinine Ratio at Week 144
Description: Urine RBP is a renal biomarker which is used to detect drug-induced kidney injury.
Time Frame: Baseline; Week 144
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 381 | 355
percent change | 37.4 [-6.0 to 87.3] | 106.9 [38.0 to 254.9]

22. Secondary Outcome: Percent Change From Baseline in Urine Beta-2-microglobulin to Creatinine Ratio at Week 48
Description: Urine Beta-2-microglobulin is a renal biomarker which is used to detect drug-induced kidney injury.
Time Frame: Baseline; Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 407 | 397
percent change | -32.8 [-58.7 to 1.3] | 18.0 [-28.8 to 171.6]

23. Secondary Outcome: Percent Change From Baseline in Urine Beta-2-microglobulin to Creatinine Ratio at Week 96
Description: Urine Beta-2-microglobulin is a renal biomarker which is used to detect drug-induced kidney injury.
Time Frame: Baseline; Week 96
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 390 | 378
percent change | -33.5 [-60.0 to 2.0] | 32.5 [-27.8 to 205.6]

24. Secondary Outcome: Percent Change From Baseline in Urine Beta-2-microglobulin to Creatinine Ratio at Week 144
Description: Urine Beta-2-microglobulin is a renal biomarker which is used to detect drug-induced kidney injury.
Time Frame: Baseline; Week 144
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 379 | 351
percent change | -24.6 [-57.5 to 13.3] | 60.4 [-10.4 to 318.8]

ADVERSE EVENTS:
Time Frame: Double-Blind Phase: Up to a maximum of 194.1 weeks plus 30 days; Open-Label Phase: Up to a maximum of 48.3 weeks plus 30 days
Description: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug.
Groups:
- Double-Blind: E/C/F/TAF: Adverse events reported in this group occurred during the Double-Blind Phase in participants who received E/C/F/TAF (150/150/200/10 mg) FDC tablet plus E/C/F/TDF placebo tablet administered orally once daily for 144 weeks.
- Double-Blind: E/C/F/TDF: Adverse events reported in this group occurred during the Double-Blind Phase in participants who received E/C/F/TDF (150/150/200/300 mg) FDC tablet plus E/C/F/TAF placebo tablet administered orally once daily for 144 weeks.
- Open-Label: E/C/F/TAF to E/C/F/TAF; Open-Label: E/C/F/TDF to E/C/F/TAF: Adverse events reported in this group occurred during the Open-Label Extension Phase in participants who switched from the Double-Blind E/C/F/TAF group to receive E/C/F/TAF (150/150/200/10 mg) FDC tablet until commercially available or until Gilead Sciences terminated the study in that country.
Arm/Group | Double-Blind: E/C/F/TAF | Double-Blind: E/C/F/TDF | Open-Label: E/C/F/TAF to E/C/F/TAF | Open-Label: E/C/F/TDF to E/C/F/TAF
Serious Adverse Events (participants affected / at risk) | 73/435 | 65/432 | 0/90 | 1/94
Other Adverse Events (participants affected / at risk) | 380/435 | 375/432 | 16/90 | 14/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind: E/C/F/TAF (N=435) | Double-Blind: E/C/F/TDF (N=432) | Open-Label: E/C/F/TAF to E/C/F/TAF (N=90) | Open-Label: E/C/F/TDF to E/C/F/TAF (N=94)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0
Incarcerated hernia (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 | 1 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 0
Acute hepatitis C (Infections and infestations) | 2 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 8 | 3 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0 | 0
Atypical mycobacterial lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Campylobacter infection (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 3 | 0 | 0
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 1 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 1 | 0 | 0
Eye infection syphilitic (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0 | 0
Hepatitis syphilitic (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 1 | 0 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 3 | 0 | 1
Meningitis viral (Infections and infestations) | 3 | 0 | 0 | 0
Mycobacterium avium complex infection (Infections and infestations) | 1 | 0 | 0 | 0
Neurosyphilis (Infections and infestations) | 0 | 1 | 0 | 0
Penile abscess (Infections and infestations) | 0 | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Psoas abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Secondary syphilis (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Shigella infection (Infections and infestations) | 0 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 2 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Kidney contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Liver contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Stab wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Uterine perforation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Prognathism (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Retrognathia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Vascular headache (Nervous system disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Drug use disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Homicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 1 | 0 | 0
Schizoaffective disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Substance use disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Substance-induced mood disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 4 | 2 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 0 | 0
Post infection glomerulonephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Scrotal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Alcohol detoxification (Surgical and medical procedures) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind: E/C/F/TAF (N=435) | Double-Blind: E/C/F/TDF (N=432) | Open-Label: E/C/F/TAF to E/C/F/TAF (N=90) | Open-Label: E/C/F/TDF to E/C/F/TAF (N=94)
Abdominal pain (Gastrointestinal disorders) | 30 | 24 | 0 | 0
Constipation (Gastrointestinal disorders) | 15 | 23 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 112 | 105 | 1 | 1
Flatulence (Gastrointestinal disorders) | 18 | 29 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 23 | 20 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 20 | 23 | 0 | 1
Nausea (Gastrointestinal disorders) | 73 | 84 | 2 | 0
Vomiting (Gastrointestinal disorders) | 39 | 26 | 0 | 0
Fatigue (General disorders) | 49 | 47 | 0 | 0
Pyrexia (General disorders) | 29 | 31 | 0 | 1
Bronchitis (Infections and infestations) | 41 | 29 | 0 | 1
Chlamydial infection (Infections and infestations) | 19 | 22 | 0 | 0
Folliculitis (Infections and infestations) | 26 | 14 | 0 | 0
Gastroenteritis (Infections and infestations) | 28 | 25 | 0 | 1
Gonorrhoea (Infections and infestations) | 22 | 20 | 0 | 2
Influenza (Infections and infestations) | 28 | 32 | 0 | 0
Pharyngitis (Infections and infestations) | 26 | 23 | 1 | 1
Sinusitis (Infections and infestations) | 43 | 25 | 0 | 0
Syphilis (Infections and infestations) | 55 | 56 | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 92 | 95 | 3 | 2
Viral upper respiratory tract infection (Infections and infestations) | 69 | 64 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 46 | 36 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 50 | 61 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 41 | 57 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 34 | 26 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 29 | 29 | 0 | 0
Dizziness (Nervous system disorders) | 30 | 25 | 0 | 0
Headache (Nervous system disorders) | 69 | 63 | 0 | 0
Anxiety (Psychiatric disorders) | 32 | 25 | 0 | 0
Depression (Psychiatric disorders) | 37 | 35 | 0 | 0
Insomnia (Psychiatric disorders) | 45 | 35 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 58 | 56 | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 34 | 25 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 24 | 9 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 37 | 27 | 1 | 0
Hypertension (Vascular disorders) | 23 | 23 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years